CLINICAL TRIAL: NCT04555980
Title: Will Warm Patch on the Injecting Site Decrease the Injection Pain Induced by Propofol
Brief Title: Warm Patch Decrease Propofol Injection Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: First People's Hospital of Chenzhou (Other)
Responsible Party: Principal Investigator, zhiming zhang, Director of Department of Anesthesiology, First People's Hospital of Chenzhou
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 202001
Record Dates: First submitted 2020-09-08; First posted 2020-09-21 (Actual); Last update posted 2020-09-21 (Actual); Status verified 2020-09

CONDITIONS: Pain Syndrome; Propofol Infusion Syndrome; Injection Site Irritation
Keywords: propofol,injection,pain
MeSH Terms: conditions — Somatoform Disorders; Propofol Infusion Syndrome

STUDY DESIGN:
Intervention Model Description: Group W : the injection site was covered with warm patch. Group C: the injection site was covered with Cotton patch.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The assessor did not know the grouping of the pain scores in memory, nor did he know the purpose of the warming patch.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Warm patch (Experimental): the injection site was covered with warm patch.
  Interventions: Device: Warming patch
- Cotton patch (Placebo Comparator): the injection site was covered with cotton patch.
  Interventions: Device: Cotton patch

INTERVENTIONS:
Device: Warming patch — The warming patch can increase the temp of injection site, result in a blood vessels to dilate, which may have some contribute to decreasing injection pain.
  Arms: Warm patch
Device: Cotton patch — The Cotton patch will cover the injection site as placebo. It dose not have the function of heating comparing to Warming patch.
  Arms: Cotton patch

SUMMARY:
Propofol causes injection pain is still a common clinical unsolved problem. Mixing a small amount of lidocaine with propofol or injecting lidocaine in advance can reduce the pain caused by propofol injection. Using an air warmer to warm the arm can also reduce the pain caused by propofol injection. Investors suspect that treatment with a warming patch (covering the injection site) can also reduce the pain caused by propofol injection.

DETAILED DESCRIPTION:
This is a single-center randomized controlled clinical study. Purpose of this study is to explore whether the coverage of the warming patch (for 5min before injection) can reduce the pain induced by propofol injection.

The patients included in the study were randomly divided into two groups. The group W used a warming patch to cover the injection site, and the group C used a cotton pad to cover the injection site. After 5 minutes of coverage, the propofol injection was induced, and the patient's complaint of pain (calling or arm withdrawal) during propofol injection was observed, and the patient's recall of the pain score during induction after the patient recovered. After the patients regained consciousness, the data of the two groups were compared to determine whether the use of the warming patch could reduce the pain caused by propofol injection.

ELIGIBILITY:
Inclusion Criteria:

* No peripheral phlebitis
* No history of Raynaud's syndrome
* No history of smoking or alcoholism
* Body mass index BMI<28 kg/cm2

Exclusion Criteria:

* Refusal of anesthesia
* Previous injection pain caused by propofol
* Difficulty in exposing the veins on the back of the hand or difficulty in venipuncture
* Complained of pain after normal saline infusion.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2020-03-20 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-06 (Actual)

PRIMARY OUTCOMES:
Arm withdrawn | 5min
  When propofol was injected, the arm was withdrawn due to injection pain.
Complaints of pain | 5min
  The patient complained about the pain of the propofol injection
Pain score after awakening from propofol | 10min
  Let the patients give a score when they recoved from propofol induced anesthesia.

SECONDARY OUTCOMES:
Respiratory depression | 5min
  those ases when pulse oxygen saturation is less than 90%
Temperature of injection site after injecting of propofol. | 10min
  Get the temperature of the back of the hand with an infrared thermometer

CONTACTS AND LOCATIONS:
Locations (1):
- Zhiming Zhang, Chenzhou, Hunan, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 180 days

REFERENCES:
- [Background] Jeong M, Yoon H. Comparison of the effects of lidocaine pre-administration and local warming of the intravenous access site on propofol injection pain: Randomized, double-blind controlled trial. Int J Nurs Stud. 2016 Sep;61:209-18. doi: 10.1016/j.ijnurstu.2016.06.012. Epub 2016 Jun 24. PMID 27372434
- [Background] Euasobhon P, Dej-Arkom S, Siriussawakul A, Muangman S, Sriraj W, Pattanittum P, Lumbiganon P. Lidocaine for reducing propofol-induced pain on induction of anaesthesia in adults. Cochrane Database Syst Rev. 2016 Feb 18;2(2):CD007874. doi: 10.1002/14651858.CD007874.pub2. PMID 26888026
- [Background] Lang BC, Yang CS, Zhang LL, Zhang WS, Fu YZ. Efficacy of lidocaine on preventing incidence and severity of pain associated with propofol using in pediatric patients: A PRISMA-compliant meta-analysis of randomized controlled trials. Medicine (Baltimore). 2017 Mar;96(11):e6320. doi: 10.1097/MD.0000000000006320. PMID 28296748